CLINICAL TRIAL: NCT02755324
Title: Establishing a Single-sex Controlled Human Schistosomiasis Infection Model: Safety and Dose Finding
Brief Title: Single-sex Controlled Human Schistosomiasis Infection: Safety and Dose Finding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, MD, PhD, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CoHSI1
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Schistosomiasis; Schistosoma Mansoni
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Volunteers will be exposed to escalating doses of male Schistosoma mansoni cercariae
  Interventions: Biological: male Schistosoma mansoni cercariae

INTERVENTIONS:
Biological: male Schistosoma mansoni cercariae — Viable male Schistosoma mansoni cercariae of the Puerto Rican strain

SUMMARY:
Groups of 3 or 7 volunteers will be exposed to a predetermined number of male Schistosoma mansoni cercariae until 10 volunteers are found infected.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 and ≤ 45 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator, is available to attend all study visits.
4. Subject will remain within Europe (excluding Corsica) during the study period and is reachable by mobile telephone from week 3 to week 12 of the study period.
5. Subject agrees to refrain from blood donation throughout the study period.
6. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
7. Subject has signed informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   * body weight <50 kg or Body Mass Index (BMI) <18.0 or >30.0 kg/m2 at screening;
   * positive HIV, hepatitis B or hepatitis C screening tests;
   * the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period;
   * history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years;
   * any history of treatment for severe psychiatric disease by a psychiatrist in the past year;
   * history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
   * Any clinically significant abnormalities (including extended QT interval) on electrocardiogram
2. The chronic use of any drug known to interact with praziquantel, or artesunate or lumefantrine metabolism (e.g. phenytoin, carbamazepine, phenobarbital, primidon, dexamethasone, rifampicin, cimetidine, flecainide, metoprolol, imipramine, amitriptyline, clomipramine, class I and III anti-arrythmics, antipsychotics, antidepressants, macrolides, fluoroquinolones, imidazole- and triazole antimycotics, antihistamines) Because lumefantrine may cause extension of QT-time, chronic use of drugs with effect on QT interval are excluded from the study.
3. For female subjects: positive urine pregnancy test at screening.
4. Any history of schistosomiasis or treatment for schistosomiasis.
5. Positive serology for schistosomiasis or elevated serum or urine circulating anodic antigen or positive Schistosoma serology at baseline.
6. Known hypersensitivity to or contra-indications (including co-medication) for use of praziquantel or, artesunate or lumefantrine.
7. Being an employee or student of the department of parasitology or infectious diseases of the Leiden University Medical Center.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Number of grade 3 and 4 adverse events, possibly, probably or definitely related to controlled human Schistosoma mansoni infection with male cercariae. | 20 weeks
The number of male cercariae at which 100% volunteers show detectable Schistosoma mansoni circulating anodic antigen (CAA). | 12 weeks

SECONDARY OUTCOMES:
Average number of weeks until positive serum circulating anodic antigen test | 12 weeks
Comparison of the height of the peak serum circulating anodic antigen concentration in low dose compared with high dose group | 12 weeks
Comparison of the humoral (antibody) response profile by protein and glycan array between infected and uninfected individuals | 1 year
Differences in in ex vivo lymphocyte profiles between infected and uninfected individuals | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Langenberg MCC, Hoogerwerf MA, Janse JJ, van Lieshout L, Corstjens PLAM, Roestenberg M; CoHSI clinical trial team. Katayama Syndrome Without Schistosoma mansoni Eggs. Ann Intern Med. 2019 May 21;170(10):732-733. doi: 10.7326/L18-0438. Epub 2019 Jan 8. No abstract available. PMID 30615787
- [Result] Langenberg MCC, Hoogerwerf MA, Koopman JPR, Janse JJ, Kos-van Oosterhoud J, Feijt C, Jochems SP, de Dood CJ, van Schuijlenburg R, Ozir-Fazalalikhan A, Manurung MD, Sartono E, van der Beek MT, Winkel BMF, Verbeek-Menken PH, Stam KA, van Leeuwen FWB, Meij P, van Diepen A, van Lieshout L, van Dam GJ, Corstjens PLAM, Hokke CH, Yazdanbakhsh M, Visser LG, Roestenberg M. A controlled human Schistosoma mansoni infection model to advance novel drugs, vaccines and diagnostics. Nat Med. 2020 Mar;26(3):326-332. doi: 10.1038/s41591-020-0759-x. Epub 2020 Feb 17. PMID 32066978